CLINICAL TRIAL: NCT03310944
Title: An Open-label, Randomized, Single-dose, 4-period, 4-sequence Crossover Relative Bioavailability Study Comparing Sotagliflozin Prototypes Tablets With Reference Tablet in Healthy Subjects
Brief Title: Comparison of Sotagliflozin Prototype Tablets With Reference Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BDR14994; 2017-002104-27; U1111-1195-6292 (Other: UTN)
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sotagliflozin dose 1 (reference formulation) (Active Comparator): Single oral dose on Day 1 of one of the four period in fasting condition
  Interventions: Drug: sotagliflozin (SAR439954)
- Sotagliflozin dose 2 (prototype p1 formulation) (Experimental): Single oral dose on Day 1 of one of the four period in fasting condition
  Interventions: Drug: sotagliflozin (SAR439954)
- Sotagliflozin dose 3 (prototype p2 formulation) (Experimental): Single oral dose on Day 1 of one of the four period in fasting condition
  Interventions: Drug: sotagliflozin (SAR439954)
- Sotagliflozin dose 4 (prototype p3 formulation) (Experimental): Single oral dose on Day 1 of one of the four period in fasting condition
  Interventions: Drug: sotagliflozin (SAR439954)

INTERVENTIONS:
Drug: sotagliflozin (SAR439954) — Pharmaceutical form: tablets
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the relative bioavailability of sotagliflozin following single doses of 3 sotagliflozin prototype tablet formulations p1, p2 and p3 versus the reference tablet formulation in fasted conditions in healthy subjects.

Secondary Objectives:

* To assess the pharmacokinetic characteristics of sotagliflozin and its 3-O-glucuronide following single doses of 3 sotagliflozin prototype tablet formulations p1, p2 and p3 and of the reference formulation in fasted conditions in healthy subjects.
* To assess the clinical and laboratory safety of single oral doses of 3 sotagliflozin prototype tablet formulations p1, p2 and p3 and the reference tablet formulation in fasted conditions in healthy subjects.

DETAILED DESCRIPTION:
Total duration is 37 to 75 days for each subject, with 2 to 21 days screening period; 4 dosing days, i.e. one in each of the 4 treatment periods. Observation period in each treatment period is 6 days. Washout between dosing days is 7 to 10 days. Follow-up visit is 14-21 days after last dosing.

ELIGIBILITY:
Inclusion criteria :

* Healthy male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 32.0 kg/m², inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position:
* 95 mmHg <systolic blood pressure (SBP) <140 mmHg,
* 45 mmHg <diastolic blood pressure (DBP) <90 mmHg,
* 40 bpm <heart rate (HR) <100 bpm.
* Standard 12-lead electrocardiogram parameters after 10 minutes resting in supine position in the following ranges; 120 ms<PR<220 ms, QRS<120 ms, QTc≤430 ms if male and QTc≤450 ms if female with normal electrocardiogram (ECG) tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and international normalized ratio (INR) should not exceed the upper laboratory norm. Activated partial thromboplastin time (aPTT) should not exceed normal control more than 10 seconds. Total bilirubin out of normal range can be acceptable if total bilirubin should not exceed 1.5 the upper limit with normal conjugated bilirubin values (unless the subject has documented Gilbert syndrome).
* Female subject must use a double contraception method including a highly effective method of birth control except if she has undergone sterilization at least 3 months earlier or is postmenopausal. The accepted double contraception methods include the use of 1 of the following contraceptive options: (1) intrauterine device; (2) condom or diaphragm or cervical/vault cap, in addition to spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma follicle-stimulating hormone (FSH) level >30 IU/L. Hormonal contraception is NOT acceptable in this study due to drug interaction.
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom) plus (spermicide or intra-uterine device or hormonal contraceptive) from the inclusion up to 4 months after the last dosing.
* Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 4 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 4 months after the last dosing.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* History of renal disease, or significant abnormal kidney function test with glomerular filtration rate (GFR) <90 mL/min as calculated using the Cockcroft-Gault equation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day)
* If female, pregnancy (defined as positive β-HCG blood test if applicable), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

Any oral contraceptives during the screening period or for at least 15 days prior to inclusion; any injectable contraceptives or hormonal intrauterine devices within 12 months prior to inclusion; or topical controlled delivery contraceptives (patch) for 3 months prior to inclusion.

* Any subject in the exclusion period of a previous study according to applicable regulations.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency Virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol test.
* Any consumption of citrus (grapefruit, orange, etc) or their juices within 5 days before inclusion.
* Any history or presence of deep leg vein thrombosis or embolism or a recurrent or frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children).
* Any presence or history of urinary tract infection or genital mycotic infection in the last 4 weeks before screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Pharmacokinetic (PK) Parameter: AUC | From 0 to 144 hours after IMP intake
  Sotagliflozin: Area under the concentration-time curve from 0 to infinity (AUC) for reference, p1, p2, and p3 formulations
Assessment of PK Parameter: Area under the concentration-time curve from 0 to last quantifiable concentration (AUClast) | From 0 to 144 hours after IMP intake
  Sotagliflozin: Area under the concentration-time curve from 0 to last quantifiable concentration for reference, p1, p2, and p3 formulations
Assessment of PK Parameter: Maximum plasma concentration (Cmax) | From 0 to 144 hours after IMP intake
  Sotagliflozin: Maximum plasma concentration (Cmax) for reference, p1, p2, and p3 formulations

SECONDARY OUTCOMES:
Assessment of PK Parameter: Tmax | From 0 to 144 hours after investigational medicinal product (IMP) intake
  Sotagliflozin: Time to reach maximum plasma concentration (Tmax)
Assessment of PK Parameter: Time to reach AUClast (Tlast) | From 0 to 144 hours after IMP intake
  Sotagliflozin: Time to reach AUClast
Assessment of PK Parameter: Terminal elimination half-life (t1/2) | From 0 to 144 hours after IMP intake
  Sotagliflozin: Terminal elimination half-life (t1/2)
Assessment of PK Parameter: Tmax | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: Tmax
Assessment of PK Parameter: Tlast | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: Time to reach AUClast
Assessment of PK Parameter: t1/2 | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: t1/2
Assessment of PK Parameter: Cmax | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: Cmax
Assessment of PK Parameter: AUC | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: AUC
Assessment of PK Parameter: AUClast | From 0 to 144 hours after IMP intake
  Sotagliflozin 3-O-glucuronide: AUClast
Adverse Events | Up to 75 days
  Number of patients with treatment emergent adverse events (serious and non-serious)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org